CLINICAL TRIAL: NCT04842279
Title: FACE-Q Measurement of the Patient Perspective in Facial Reconstructive Surgery: A Prospective Database
Brief Title: FACE-Q in Facial Reconstructive Surgery: A Prospective Database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mark McRae, Principal Investigator, McMaster University
Other Study IDs: 9446
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Skin Cancer, Basal Cell Skin Cancer Skin Cancer, Non-Melanoma Skin Cancers - Squamous Cell Carcinoma Patient Satisfaction
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FACE-Q scale — FACE-Q is a recently developed and validated patient reported outcome measure (PROM) tool that allows clinicians to assess patient perspectives after skin cancer surgery of the face.The PROM is used to assess the perspective and impact of skin cancer as well as its treatment on the patient's quality of life (QoL). Patients with skin cancer may have increased anxiety, social isolation, and cosmetic concerns after surgery. The FACE-Q utilizes five scales to measure the psychometric, QoL, patient experience, and cosmetic outcomes. Raw scores are transformed to a 0-100 scale with a higher score indicating a better outcome.
  Any studies using FACE-Q for facial surgery reconstruction at our center may be eligible for inclusion in the database

SUMMARY:
The primary objective is to establish a prospective database of clinical information, FACE-Q scores, and patient photographs (as appropriate) to enhance the understanding and practice of facial plastic and reconstructive surgery.

DETAILED DESCRIPTION:
Patient perspective is essential as medicine progresses to become more patient centered. FACE-Q is a recently developed and validated patient-reported outcome measure (PROM) tool that allows clinicians to assess patient perspectives after skin cancer surgery of the face. The FACE-Q has more than 40 independent scales and checklist each measuring different patient reported outcomes (PRO).

The FACE-Q utilizes five scales to measure the psychometric, QoL, patient experience, and cosmetic outcomes. The FACE-Q was validated in both surgical and non-surgical patients. This is a single-center project to establish a prospective database of clinical information from patients who utilize FACE-Q in a clinical investigation. This database is being established in efforts to promote research in various patient populations Rationale The purpose of this prospective database would be to evaluate levels of satisfaction and QoL across various interventions and patient populations after using the FACE-Q PROM. Long term data collection will include information related to QoL, patient experience, and cosmetic outcomes. Many areas related to patient reported outcomes in the context of facial reconstruction surgery are in their early years. There are many areas of research needed to aid in clinical decision making. The database will allow these questions to be answered using a retrospective model and will provide the background information required to mount larger scale randomized controlled trials, when possible. Information collected in the database will also allow meaningful research to be conducted in a timely and cost-effective manner. For example database information could help answer, "Which patient characteristics are associated with higher FACE-Q scores in non-melanoma facial cancer patients?". The investigators will initiate a line of investigations that will characterize adults who use the FACE-Q in various clinical contexts with the ultimate goal of improving patient outcomes.

The study was designed in concordance with the Enhancing the Quality and Transparency of Health Research (EQUATOR) reporting guidelines using: The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE), and Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) statements as well as based off previous prospective studies that used FACE-Q for PROMs.

ELIGIBILITY:
Inclusion Criteria:

i. Age 18 years or older ii. Use of any module of the FACE-Q scale to measure a patient-reported outcome iii. Ability to provide informed consent

Exclusion Criteria:

i. Those patients who do not meet all of the above inclusion criteria will be excluded from the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This database will collect existing or prospective data that is part of standard clinical care from the electronic medical record of patients which are part of any FACE-Q studies.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-20 (Estimated); Primary Completion 2021-07-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
FACE-Q score | 12 months
  FACE-Q is a recently developed and validated patient reported outcome measure (PROM) tool that allows clinicians to assess patient perspectives after skin cancer surgery of the face.The PROM is used to assess the perspective and impact of skin cancer as well as its treatment on the patient's quality of life (QoL). Patients with skin cancer may have increased anxiety, social isolation, and cosmetic concerns after surgery. The FACE-Q utilizes five scales to measure the psychometric, QoL, patient experience, and cosmetic outcomes. Raw scores are transformed to a 0-100 scale with a higher score indicating a better outcome

SECONDARY OUTCOMES:
Facial photos | 12 months
  Patient photos may be taken post-op from the other studies and will be included if performed

CONTACTS AND LOCATIONS:
Overall Officials: Mark McRae, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huynh MNQ, Olaiya O, Kim PJ, Gallo L, Dunn E, Farrokhyar F, McRae MC, Voineskos S, McRae MH. A comparison of skin grafts versus local flaps for facial skin cancer from the patient perspective: protocol for a feasibility study. Jpn J Clin Oncol. 2023 Jun 1;53(6):489-493. doi: 10.1093/jjco/hyad018. PMID 36946321